CLINICAL TRIAL: NCT06176469
Title: Population-level Prevalence, Effect on Quality of Life, and Treatment Behavior for Renal Colic and Urolithiasis in Poland
Brief Title: Renal Colic and Urolithiasis in Poland
Acronym: POLSTONE
Status: Active, not recruiting | Type: Observational
Sponsor: Mikolaj Przydacz (Other)
Responsible Party: Sponsor-Investigator, Mikolaj Przydacz, Associate Professor, Jagiellonian University
Organization: Jagiellonian University (Other)
Other Study IDs: 118.6120.94.2023
Record Dates: First submitted 2023-12-09; First posted 2023-12-19 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Renal Colic; Urolithiasis
MeSH Terms: conditions — Renal Colic; Urolithiasis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Population-level and representative cohort
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The aim of this study is to analyze the prevalence, effect on quality of life, and treatment-related behaviors for renal colic and urolithiasis in a population-representative sample of Poles. We will be using an Internet interview format for renal colic and urolithiasis evaluation. The study will include respondents representative for age and place of residence with adequate proportions of respondents from urban and rural areas.

ELIGIBILITY:
Inclusion Criteria:

- consent to participate

Exclusion Criteria:

- lack of consent to participate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A representative pool of men and women in Poland
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of renal colic and urolithiasis in Poland | December 2023 - December 2024
  Prevalence of renal colic and urolithiasis in Poland

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Jagiellonian University, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT06176469/Prot_000.pdf